CLINICAL TRIAL: NCT04275414
Title: Effecacy and Safety of Bevacizumab in Severe Patients With Covid-19: a Pilot Study (BEST-CP)
Brief Title: Bevacizumab in Severe or Critical Patients With COVID-19 Pneumonia
Acronym: BEST-CP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: Renmin Hospital of Wuhan University (Other); Moriggia-Pelascini Gravedona Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QLEmer20200214
Record Dates: First submitted 2020-02-14; First posted 2020-02-19 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-02

CONDITIONS: Coronavirus Infections
Keywords: COVID-19; Bevacizumab; pneumonia
MeSH Terms: conditions — Coronavirus Infections; COVID-19; Pneumonia | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- bevacizumab plus standard care (Experimental): Under ECG monitoring, give bevacizumab 500mg + 0.9% sodium chloride solution 100ml via intravenous drip, time is no less than 90min.
  Interventions: Drug: Bevacizumab Injection

INTERVENTIONS:
Drug: Bevacizumab Injection — Bevacizumab 500mg + normal saline (NS) 100ml, ivdrip ≥90min

SUMMARY:
The novel identified coronavirus (SARS-CoV-2) in 2019 causes an nationwide outbreak as well as public health crisis in China, and expands globally. Pulmonary edema is one of the most detrimental symptoms and usually presents in severe and critical coronavirus disease (COVID-19), resulting in dyspnea, acute lung injury (ALI) ,acute respiratory distress syndrome (ARDS), and even death. Recent evidence revealed higher levels of blood Vascular Endothelial Growth Factor (VEGF) in COVID-19 patients compared with healthy controls. VEGF is considered as the most potent vascular permeability inducers. Numerous studies have revealed that VEGF was a key factor and a potential therapeutic target in ALI and ARDS. Bevacizumab, an anti-VEGF drug, approved by the FDA on February 26, 2004 and widely used in clinical oncotherapy, is a promising drug for ALI/ARDS in COVID-19 through suppression of pulmonary edema.

DETAILED DESCRIPTION:
In December 2019, a new identified coronavirus (SARS-CoV-2) outbreak in Wuhan, causes public health crisis in China and spreads worldwide. On February 11,2020, the World Health Organization officially named the disease caused by the new coronavirus "COVID-19". The Chinese Government takes stronger and harsher measures to control the progression of its outbreak. Meanwhile, five editions of "Diagnosis and Treatment for Novel Coronavirus-Infected Pneumonia" has been timely and continuously issued, which play extremely important roles in guiding the clinical management of COVID-19 nationwide in China.

The symptoms of human infection with SARS-CoV-2 are generally fever, fatigue, dry cough and dyspnea. Noteworthy, a considerable percentage of COVID-19 cases have rapidly progressed to severe and critical type, among which acute lung injury (ALI) and acute respiratory distress syndrome (ARDS) are the most common complications, resulting in a large number of pneumonia hospitalized patients requiring supplemental oxygen, mechanical ventilation, or even ECMO.Pulmonary edema is a detrimental feature as well as a key causal factor of ALI/ARDS.

Vascular Endothelial Growth Factor (VEGF) is considered as the most potent vascular permeability inducers. Recent evidence has revealed higher VEGF levels in COVID-19 patients compared with healthy controls. The rise of VEGF levels may be caused by hypoxia, severe inflammation, and upregulation of the infected respiratory tract epithelium itself. Numerous studies have confirmed a key role of VEGF as potential therapeutic target in acute lung injury (ALI) and acute respiratory distress syndrome (ARDS) due do increase vascular permeability and induce pulmonary edema.

Thus, Bevacizumab, an anti-VEGF medication, may offer a unique approach to treat ALI/ARDS caused by COVID-19. Bevacizumab is a humanized monoclonal antibody with long half-life. It has been approved by the FDA on February 26, 2004 and widely used in clinical oncotherapy, with the pharmacokinetics and pharmacodynamics having been widely understood. Therefore, Bevacizumab is a promising drug for the treatment of ALI/ARDS as well as reduction of mortality in severe and critical COVID-19 patients through suppression of pulmonary edema.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 80.
2. Confirmed COVID-19 diagnosis(including the clinically confirmed cases in Hubei).
3. Accord with any of the following: respiratory distress, RR ≥ 30 breaths/min; or SpO2 ≤ 93% at rest; or partial arterial oxygen pressure (PaO2) / fraction of inspiration O2 (FiO2) >100mmHg and ≤ 300mmHg (1mmHg = 0.133kPa).
4. Chest imaging confirms lung involvement and has inflammatory exudation or pleural effusion.

Exclusion Criteria:

1. Cannot obtain informed consent.
2. Severe hepatic dysfunction (Child Pugh score ≥ C, or AST> 5 times the upper limit); Severe renal dysfunction (estimated glomerular filtration rate ≤ 30mL / min / 1.73 m2) or receive continuous renal replacement therapy, hemodialysis, or peritoneal dialysis.
3. Unsatisfactory controlled hypertension (seated systolic blood pressure> 160mmHg, or diastolic blood pressure> 100mmHg); previous history of hypertension crisis or hypertensive encephalopathy.
4. Poorly controlled heart diseases, such as NYHA class II and above cardiac insufficiency, unstable angina pectoris, myocardial infarction within 1 year before enrollment, supraventricular or ventricular arrhythmia need treatment or intervention.
5. Hereditary bleeding tendency or coagulopathy; received full-dose anticoagulant or thrombolytic therapy within10 days before enrollment, or have taken non-steroidal anti-inflammatory drugs with platelet suppression within 10 days before enrollment (Except those who use small doses of aspirin ≤325mg / day for preventive use).
6. Thrombosis within 6 months before enrollment. And from those patients, screen who had arterial / venous thromboembolic events, such as, ischemic stroke, transient ischemic attack, deep venous thrombosis, pulmonary embolism, etc. within 1 year ahead of enrollment. Severe vascular disease (including aneurysms or arterial thrombosis requiring surgery) within 6 months before enrollment.
7. Unhealed wounds, active gastric ulcers or fractures. Gastrointestinal perforation, gastrointestinal fistula, abdominal abscess, visceral fistula formation within 6 months before enrollment. Major surgery (including preoperative Chest biopsy) or major trauma (such as a fracture) within 28 days before enrollment. May have surgery during the trial.
8. Severe, active bleeding such as hemoptysis, gastrointestinal bleeding, central nervous system bleeding, and nosebleeds within 1 month before enrollment.
9. Malignant tumors within 5 years before enrollment.
10. Allergic to bevacizumab or its components.
11. Untreated active hepatitis or HIV-positive patients.
12. Pregnant and lactating women and those planning to get pregnant.
13. Participated in other clinical trials, not considered suitable for this study by the researchers.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-02-15 (Actual); Primary Completion 2020-04-05 (Actual); Study Completion 2020-05-02 (Actual)

PRIMARY OUTCOMES:
Partial arterial oxygen pressure (PaO2) to fraction of inspiration O2 (FiO2) ratio | 24 hours
  Partial arterial oxygen pressure (PaO2) to fraction of inspiration O2 (FiO2) ratio
Partial arterial oxygen pressure (PaO2) to fraction of inspiration O2 (FiO2) ratio | 7 days
  Partial arterial oxygen pressure (PaO2) to fraction of inspiration O2 (FiO2) ratio

SECONDARY OUTCOMES:
Rate of improvement of oxygen-support status | 28 days
  The oxygen-support status includes 6 levels: mechanical ventilation, non-invasive ventilation, a transition status of alternate use of non-invasive ventilation and high-flow oxygen, high-flow oxygen, low-flow oxygen and ambient air. The improvement of oxygen-support status is defined as switch from a higher level of oxygen-support to a lower level.
The change of areas of pulmonary lesions shown on chest radiological imaging (chest CT or X-ray) | 7 days
  The areas of pulmonary lesions are analysised by a professional imaging software.
Blood lymphocyte counts | 7 days
  Blood lymphocyte counts
Level of CRP | 7 days
  Level of CRP
Level of hs-CRP | 7 days
  Level of hs-CRP
All-cause mortality | 28 days
  All-cause mortality
Discharge rate | 28 days
  Discharge rate

CONTACTS AND LOCATIONS:
Overall Officials: Yuguo Chen, Dr, Principal Investigator — Qilu Hospital of Shandong University
Locations (3):
- China (2):
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Qilu Hospital of Shandong University, Jinan, Shandong
- Moriggia-Pelascini Gravedona Hospital, Gravedona, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pang J, Xu F, Aondio G, Li Y, Fumagalli A, Lu M, Valmadre G, Wei J, Bian Y, Canesi M, Damiani G, Zhang Y, Yu D, Chen J, Ji X, Sui W, Wang B, Wu S, Kovacs A, Revera M, Wang H, Jing X, Zhang Y, Chen Y, Cao Y. Efficacy and tolerability of bevacizumab in patients with severe Covid-19. Nat Commun. 2021 Feb 5;12(1):814. doi: 10.1038/s41467-021-21085-8. PMID 33547300